CLINICAL TRIAL: NCT07304284
Title: Phase I/III, Multicenter, Observer-Blinded, Randomized, Active Controlled Trial to Evaluate Immunogenicity Non-Inferiority, Safety and Lot-to-Lot Consistency of Biovac OCV-S to Euvichol®-Plus in 1 to 45 Years Old South Africans
Brief Title: Trial to Evaluate Immunogenicity Non-Inferiority, Safety and Lot-to-Lot Consistency of Biovac OCV-S to Euvichol®-Plus
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: BioVac (Unknown); Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVI BIOVAC OCV-S 001
Record Dates: First submitted 2025-12-11; First posted 2025-12-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cholera Vaccination
Keywords: Biovac OCV-S; Euvichol®-Plus; IVI BIOVAC OCV-S 001; International Vaccine Institute (IVI); Biovac Institute; South African Medical Research Council (SAMRC)
MeSH Terms: interventions — Cholera Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Arm A1: Biovac OCV-S (Experimental): Biovac OCV-S (Lot 1), HIV Negative Group, 18-45 years
  Interventions: Biological: Experimental: Biovac OCV-S (inactivated whole-cell monovalent (O1) oral cholera vaccine)
- Arm A2: Biovac OCV-S (Experimental): Biovac OCV-S (Lot 2), HIV Negative Group, 18-45 years
  Interventions: Biological: Experimental: Biovac OCV-S (inactivated whole-cell monovalent (O1) oral cholera vaccine)
- Arm A3: Biovac OCV-S (Experimental): Biovac OCV-S (Lot 3), HIV Negative Group, 18-45 years
  Interventions: Biological: Experimental: Biovac OCV-S (inactivated whole-cell monovalent (O1) oral cholera vaccine)
- Arm A4: Euvichol®-Plus (Active Comparator): Euvichol®-Plus, HIV Negative Group, 18-45 years
  Interventions: Biological: Active Comparator, Euvichol®-Plus
- Arm B1: Biovac OCV-S (Experimental): Biovac OCV-S, HIV Negative Group, 6-17 years
  Interventions: Biological: Experimental: Biovac OCV-S (inactivated whole-cell monovalent (O1) oral cholera vaccine)
- Arm B2: Euvichol®-Plus (Active Comparator): Euvichol®-Plus, HIV Negative Group, 6-17 years
  Interventions: Biological: Active Comparator, Euvichol®-Plus
- Arm C1: Biovac OCV-S (Experimental): Biovac OCV-S, HIV Negative Group, 1-5 years
  Interventions: Biological: Experimental: Biovac OCV-S (inactivated whole-cell monovalent (O1) oral cholera vaccine)
- Arm C2: Euvichol®-Plus (Active Comparator): Euvichol®-Plus, HIV Negative Group, 1-5 years
  Interventions: Biological: Active Comparator, Euvichol®-Plus
- Arm AA1: Biovac OCV-S (Experimental): Biovac OCV-S, People living with HIV, 18-45 years
  Interventions: Biological: Experimental: Biovac OCV-S (inactivated whole-cell monovalent (O1) oral cholera vaccine)
- Arm AA2: Euvichol®-Plus (Active Comparator): Euvichol®-Plus, People living with HIV, 18-45 years
  Interventions: Biological: Active Comparator, Euvichol®-Plus

INTERVENTIONS:
Biological: Experimental: Biovac OCV-S (inactivated whole-cell monovalent (O1) oral cholera vaccine) — Two doses (1.5mL) at two weeks interval given orally.
  Arms: Arm A1: Biovac OCV-S; Arm A2: Biovac OCV-S; Arm A3: Biovac OCV-S; Arm AA1: Biovac OCV-S; Arm B1: Biovac OCV-S; Arm C1: Biovac OCV-S
Biological: Active Comparator, Euvichol®-Plus — Two doses (1.5mL) at two weeks interval given orally.
  Arms: Arm A4: Euvichol®-Plus; Arm AA2: Euvichol®-Plus; Arm B2: Euvichol®-Plus; Arm C2: Euvichol®-Plus

SUMMARY:
This Phase I/III clinical trial is intended to establish the immunogenicity and safety profile of Biovac OCV-S compared to available WHO pre-qualified vaccine Euvichol®-Plus in healthy adults and children and in adult people living with HIV (PLWH). The lot-to-lot consistency of Biovac OCV-S in healthy adults will also be determined.

DETAILED DESCRIPTION:
This is a phase I/III, multicenter, observer-blinded, age-descending, randomized, active controlled trial being conducted in South Africa to evaluate the immunogenicity non-inferiority and safety of Biovac OCV-S compared to Euvichol®-Plus among adults and children, and to evaluate the lot-to-lot consistency of Biovac OCV-S in adults.

A total of 2824 participants aged 1-45 years will be enrolled in the study in 4 cohorts: cohort A (1272 healthy adults aged 18-45 years), cohort AA (160 people living with HIV (PLWH) aged 18-45 years), cohort B (696 healthy children aged 6-17 years), and cohort C (696 healthy children aged 1-5 years). Participants in cohort A will be randomized into 4 arms to receive either one of the 3 lots of Biovac OCV-S or to receive the comparator Euvichol®-Plus in 1:1:1:1 ratio. Participants in cohorts AA, B and C will each be randomized into 2 arms to receive either Biovac OCV-S or Euvichol®-Plus in 3:1 ratio.

Each of the study participants will receive the assigned investigational product Biovac OCV-S or Euvichol®-Plus given orally in 2 doses at 2 weeks interval and will be followed up for safety and immunogenicity at specific time points. Each participant will be in the study for approximately 27 weeks.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (for healthy/HIV-negative cohorts A, B and C)

1. Healthy participants aged 1 to 45 years at consent
2. Participants/Parent(s)/Legally Authorized Representative (LAR) willing to provide informed consent/assent
3. HIV negative
4. Not pregnant or lactating

Inclusion Criteria (for PLWH (HIV-positive) cohort AA)

1. PLWH adults aged 18 to 45 years at consent
2. Participants on anti-retroviral (ARV) therapy with CD4 counts >350 and viral loads that are undetectable.
3. Not pregnant or lactating

Exclusion Criteria:

1. Known history or allergy to investigational vaccine components, other preventive vaccines, or any other allergies
2. Individuals with major congenital abnormalities
3. Known history of immune function disorders including immunodeficiency diseases (known HIV infection in healthy participant cohorts) or other immune function disorders (all cohorts).
4. Use of systemic steroids within past 6 months (>10 mg/day prednisone equivalent for periods exceeding 2 consecutive weeks), or receive chemotherapy, radiation therapy or other immunosuppressive drugs within the past 6 months.
5. Behavioral or cognitive impairment, chronic substance abuse, or psychiatric disease or neurological disorders.
6. Individuals with a known bleeding disorder.
7. Receipt of blood, blood-derived products, or immunoglobulin products in the past 3 months.
8. Individuals who have received other vaccines from 4 weeks prior to or within 4 weeks after any dose of the investigational product.
9. Individuals with active or previous Vibrio cholerae infection.
10. Individuals with receipt of a cholera vaccine in the past 5 years.

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2824 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Seroconversion of vibriocidal titers against Vibrio cholerae O1 Inaba and O1 Ogawa | 2 weeks after second dose of either Biovac OCV-S (i.e., one lot of Biovac OCV-S) or Euvichol®-Plus
  Proportion of participants showing seroconversion of vibriocidal titers against Vibrio cholerae O1 Inaba and O1 Ogawa (seroconversion is defined as at least 4-fold increase of vibriocidal titers compared to baseline) at 2 weeks after second dose of either Biovac OCV-S (i.e., one lot of Biovac OCV-S) or Euvichol®-Plus for all ages, in the HIV negative group.
Incidence of Treatment-Emergent Adverse Events in the HIV negative group | Within 14 days after each vaccination
  Safety of each investigational product dose at a specified duration in the HIV negative group:
  1. Occurrence of any Serious Adverse Event (SAE)/ Adverse Event of Special Interest (AESI)/ Medically Attended Adverse Event (MAAE) from the first dose vaccination throughout the final study visit
  2. Occurrence of immediate adverse events within 30 minutes after each dose vaccination
  3. Occurrence of solicited adverse events within 7 days after each dose vaccination
  4. Occurrence of unsolicited adverse events within 14 days after each dose vaccination

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of vibriocidal antibodies against Vibrio cholerae O1 Inaba and Ogawa for all ages | 2 weeks after second dose of either Biovac OCV-S (i.e., one lot of Biovac OCV-S) or Euvichol®-Plus
  GMT of vibriocidal antibodies against Vibrio cholerae O1 Inaba and Ogawa 2 weeks after second dose of either Biovac OCV-S (i.e., one lot of Biovac OCV-S) or Euvichol®-Plus for all ages, in the HIV negative group.
Proportion of participants showing seroconversion against Vibrio cholerae O1 Inaba and Ogawa | 2 weeks after second dose of either Biovac OCV-S (i.e., one lot of Biovac OCV-S) or Euvichol®-Plus
  The proportion of participants showing seroconversion against Vibrio cholerae O1 Inaba and Ogawa 2 weeks after second dose of either Biovac OCV-S (i.e., one lot of Biovac OCV-S) or Euvichol®-Plus in each age stratum, in the HIV negative group.
GMT of vibriocidal antibodies against Vibrio cholerae O1 Inaba and Ogawa in each age stratum | 2 weeks after second dose of either Biovac OCV-S (i.e., one lot of Biovac OCV-S) or Euvichol®-Plus
  GMT of vibriocidal antibodies against Vibrio cholerae O1 Inaba and Ogawa 2 weeks after second dose of either Biovac OCV-S (i.e., one lot of Biovac OCV-S) or Euvichol®-Plus in each age stratum, in the HIV negative group.
GMT of vibriocidal antibodies against Vibrio cholerae O1 Inaba and Ogawa in adults | 2 weeks after second dose of 3 lots of Biovac OCV-S
  GMT of vibriocidal antibodies against Vibrio cholerae O1 Inaba and Ogawa 2 weeks after second dose of 3 lots of Biovac OCV-S in adults in the HIV negative group.

OTHER OUTCOMES:
Proportion of participants showing seroconversion of vibriocidal titers against Vibrio cholerae O1 Inaba and Ogawa | 2 weeks after second dose of 3 lots of Biovac OCV-S
  The proportion of participants showing seroconversion of vibriocidal titers against Vibrio cholerae O1 Inaba and Ogawa 2 weeks after second dose of 3 lots of Biovac OCV-S in adults in the HIV negative group.
Seroconversion rate and GMT of vibriocidal antibodies | 2 weeks after first dose of either Biovac OCV-S or Euvichol®-Plus
  Seroconversion rate and GMT of vibriocidal antibodies 2 weeks after first dose of either Biovac OCV-S or Euvichol®-Plus for all ages and for each age stratum, in the HIV negative group.
Seroconversion rate and GMT of vibriocidal antibodies | 2 weeks after one and two doses of Biovac OCV-S and Euvichol®-Plus
  Seroconversion rate and GMT of vibriocidal antibodies 2 weeks after one and two doses of Biovac OCV-S and Euvichol®-Plus for adults, in the PLWH group.
Incidence of Treatment-Emergent Adverse Events in the PLWH group | Within 14 days after each dose vaccination
  Safety of each investigational product dose at a specified duration in the PLWH group:
  1. Occurrence of any SAE/AESI/MAAE from the first dose vaccination throughout the final study visit
  2. Occurrence of immediate adverse events within 30 minutes after each dose vaccination
  3. Occurrence of solicited adverse events within 7 days after each dose vaccination
  4. Occurrence of unsolicited adverse events within 14 days after each dose vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Saluja, MD, Principal Investigator — International Vaccine Institute; Glenda Gray, MD, Principal Investigator — Medical Research Council, South Africa; Julia Lynch, MD, Study Director — International Vaccine Institute
Locations (5):
- South Africa (5):
  - Synergy Biomed Research Institute, Durban, Eastern Cape
  - Perinatal HIV Research Unit (PHRU), Johannesburg, Gauteng
  - Wits Vaccines & Infectious Diseases Analytics (VIDA) Research Unit, Johannesburg, Gauteng
  - SAMRC Chatworth CRS, Durban, KwaZulu-Natal
  - SAMRC Isipingo CRS, Durban, KwaZulu-Natal

IPD SHARING:
Plan to Share IPD: No